CLINICAL TRIAL: NCT01853865
Title: Follow-up of Endometrial Cancer Patients: A Valuable Medical Intervention or a Dispensable Force of Habit?
Brief Title: Follow-up of Endometrial Cancer Patients
Acronym: OPAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: Research Unit of General Practice, Odense (Other); University of Southern Denmark (Other); Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Mette Moustgaard Mathiesen, PhD student, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OPAL
Record Dates: First submitted 2013-04-22; First posted 2013-05-15 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Endometrial Cancer
Keywords: Endometrial cancer; Follow-up examination
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Follow-up (No Intervention): Patients in this arm attend regular follow-up examinations, as is the current standard, at the department of gynecology following surgery.
- Self-referral (Experimental): Instead of regular follow-up examinations, this group is carefully instructed in alarm symptoms that require contact with a physician.
  Interventions: Other: Instruction in self-referral

INTERVENTIONS:
Other: Instruction in self-referral
  Other Names: Patient-initiated follow-up
  Arms: Self-referral

SUMMARY:
The present study is conducted, to elucidate the value of follow-up examinations in endometrial cancer patients. Specifically the objective is to compare hospital-based follow-up examinations with instruction in self-referral in stage I endometrial cancer patients.

The investigators hypothesize that the intervention, instruction in self-referral, will:

* reduce fear of recurrence
* improve quality of life
* improve cost-utility
* not affect disease-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with stage I Endometrial Cancer

Exclusion Criteria:

* Dementia or other mental/cognitive impairment
* Illiterate in Danish
* Treated with adjuvant chemo- and/or radiotherapy
* high risk histology
* grade 3
* follow-up for other gynecologic malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2013-05; Primary Completion 2017-12 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Fear of Cancer Recurrence Inventory (questionnaire) | change in score between 1, 10 and 34 months

SECONDARY OUTCOMES:
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | change in score between 1, 10 and 34 months
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Endometrial cancer Module (EORTC QLQ-EN24) | change in score between 1, 10 and 34 months
Posttraumatic Growth Inventory | change in score between 1, 10 and 34 months
EQ-5D-5L | change in score between 1, 10 and 34 months
Items on Unmet needs from the "Coherence for cancer patients questionnaire" | change in score between 1, 10 and 34 months
Disease-free survival | 3 years following treatment
Incidence of disease recurrence | 3 years following treatment
Resource use at hospital, primary care and use of medicinal products | During the three years following treatment
  Resource use at hospital: will be measured through questionnaires completed by relevant personnel.
  Information on resource use at primary care and use medicinal products: will be collected through the National Insurance Register and the Medicinal Product Register respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Mette M Mathiesen, Principal Investigator — Department of Gynecology, Odense University Hospital; Ole Mogensen, Professor, Study Chair — Department of Gynecology, Odense University Hospital; Pernille T Jensen, PhD, Study Chair — Department of Gynecology, Odense University Hospital; Dorte G Hansen, Lector, PhD, Study Chair — Research Unit of General Practice, Odense University Hospital
Locations (3):
- Denmark (3):
  - Aalborg University Hospital, Aalborg
  - Research Unit of gynecology, Odense University hospital, Odense C
  - Roskilde Hospital, Roskilde